CLINICAL TRIAL: NCT07016386
Title: Ultrasound-guided Interscalene Block (ISB) Versus Infraspinatus-Teres Minor (ITM) Interfacial Plane Block in Shoulder Arthroscopic Surgery
Brief Title: Ultrasound-guided Interscalene Block Versus Infraspinatus-Teres Minor Plane Block in Shoulder Arthroscopy
Acronym: (ISB)-(ITM)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Emad Lotfy Mohammed Ahmed, Lecturer of Anesthesia, SICU & Pain management, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022/0126
Record Dates: First submitted 2025-05-24; First posted 2025-06-11 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Pain; Pain Management; Pain Management in Postoperative Care
Keywords: Ultrasound guided,; interscaline block,; versus infraspinatus-teres minor block; shoulder arthroscopy.
MeSH Terms: conditions — Pain; Agnosia | interventions — SLC22A18 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants, care providers and outcome assessor will be blind regarding the procedure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A : Ultrasound guided Interscalene block (ISB) technique (Active Comparator): Interscalene block (ISB) technique, patients will be place in the supine position and the patient's head facing away from the side to be blocked. The Ultrasound probe will be applied in sterile fashion on the supraclavicular fossa to find the brachial plexus division lateral to the subclavian artery. Then, the probe will be traced cephalad to the C5-C6 root and interscalene muscles at the level of the cricoid cartilage
  Interventions: Procedure: Group A: will receive an ultrasound-guided interscalene block (ISB)
- Group B: Ultrasound guided Infraspinatus-teres minor (ITM) interfacial plane block technique (Experimental): Infraspinatus-teres minor (ITM) interfacial plane block technique, Patients will be placed in the lateral position, and a pillow will be wedged under the anterior shoulder and upper arm. The Ultrasound probe will be applied in sterile fashion and put angled obliquely, to be perpendicular to the direction of muscles to obtain the transverse scan of muscles for the ITM block. After palpation of the posterolateral corner of the acromion, the muscle-tendon units of infraspinatus (IS) and teres minor (Tm) on the humeral head will be identified below the corner. At this time, the probe will be moved slightly caudad to identify the borders of Tm. Once the IS and Tm on the humeral head area identified, by moving the probe medio caudally, the interfascial structure of the IS and Tm could be traced on the posterior surface area of the neck of the scapula.
  Interventions: Procedure: Group B:will receive an ultrasound-guided infraspinatus-teres minor (ITM) interfacial plane block

INTERVENTIONS:
Procedure: Group A: will receive an ultrasound-guided interscalene block (ISB) — Group A: will receive an ultrasound-guided interscalene block (ISB) using a 15ml mixture of lidocaine (7.5ml 2%) and bupivacaine (7.5ml 0.5%).
  Arms: Group A : Ultrasound guided Interscalene block (ISB) technique
Procedure: Group B:will receive an ultrasound-guided infraspinatus-teres minor (ITM) interfacial plane block — Group B:will receive an ultrasound-guided infraspinatus-teres minor (ITM) interfacial plane block using a 15ml mixture of lidocaine (7.5ml 2%) and bupivacaine (7.5ml 0.5%).
  Arms: Group B: Ultrasound guided Infraspinatus-teres minor (ITM) interfacial plane block technique

SUMMARY:
This study aims to compare the efficacy and safety of ultrasound-guided Interscalene block (ISB) versus Infraspinatus-Teres minor (ITM) interfacial plane block in shoulder arthroscopic surgery.

A prospective, randomized clinical trial will be conducted with 46 patients. Approval was obtained from the Medical Ethics Committee (2022/0126), and written informed consent will be collected from all participants. Patients aged 20-70, ASA I-II, scheduled for arthroscopic shoulder surgery will be divided before the induction of general anesthesia (GA) into two groups:

Group A: will receive the ultrasound guided ISB technique with a 15ml solution of 7.5ml lidocaine 2% and 7.5ml bupivacaine 0.5% be injected between the anterior and middle scalene muscles.

Group B: will receive the ultrasound guided ITM block with the same anesthetic solution be injected between the infraspinatus and teres minor muscles.

Researchers will examine the following outcomes;

1. Primary outcome measure: Efficacy of analgesia by Pain score; will be measured by Numerical Rating Scale (NRS) score (0=no pain,1-3=mild,4-6=moderate,7-9=sever,10=most sever) at postoperative 12 hour.
2. Secondary outcome measures:

   1. Duration of analgesia, starting from recovery from general anesthesia (GA) to 1st time giving the patient rescue analgesia ( measured by NRS pain score at 0, 6 ,12, 18 and 24 postoperative hours)
   2. Risk of complications from techniques
   3. Patient satisfaction after surgery.
   4. Rescue analgesic consumption
   5. Hemodynamics monitoring; measurements of heart rate and mean arterial blood pressure before induction of anesthesia and every 15 minutes during surgery till end of surgery

DETAILED DESCRIPTION:
I. Study design:

Randomized comparative study.

II. Study setting and location:

The study will be conducted at the operative room of Souad Kafafi University Hospital (SKUH), Misr University of science and Technology (MUST).

III. Study population:

Patients aged from 20 to 60 years old scheduled for shoulder surgery will be randomized in a 1:1 ratio after induction of general anesthesia (GA) to either: Group A: Received the ultrasound guided ISB technique with a 15ml solution of 7.5ml lidocaine 2% and 7.5ml bupivacaine 0.5% injected between the anterior and middle scalene muscles.

Group B: Received the ultrasound guided ITM block with the same anesthetic solution injected between the infraspinatus and teres minor muscles.

IV. Study procedures:

1. Randomization Patients will be randomly allocated by a computer-generated table into one of the study groups; the randomization sequence will be concealed in sealed opaque envelopes.
2. Study protocol

   * All Patients will have a pre-operative assessment visit, which will include; history taking, complete physical examination and review of all the results of the routine investigations (CBC, Coagulation profile, renal functions, liver functions).
   * On Arrival to the preparation room, they will receive the following premedication via intravenous (IV) route: Midazolam 0.03 mg/kg, Ondansetron 4 mg and Omeprazole 40 mg iv infusion.
   * Upon Arrival to the operating room, standard monitoring will be applied which include: Pulse Oximeter, Noninvasive Blood Pressure and Six-lead electrocardiogram (ECG).
   * General anesthesia will be induced using: Propofol 1-2mg/kg, Fentanyl1-2 μg/kg, Morphine 0.1mg/kg and Atracurium 0.5 mg/kg.
   * After endotracheal intubation, side way capnography will be applied to measure end tidal CO2 pressure in the expired air.
   * General anesthesia will be maintained using Sevoflurane 1-2 MAC (Mean Alveolar Concentrations) in O2/ Air 50% / 50%, Paracetamol 1gm iv infusion, ketorolac 30 mg iv and incremental doses of Atracurium 0.1mg/kg/30 minutes.

The patients will be randomly allocated into two groups:

Group A:

Ultrasound-guided Interscalene block (ISB) technique.

Group B:

Ultrasound-guided Infraspinatus-teres minor (ITM) interfacial plane block technique

V. Study outcomes:

1. Primary outcome measure:

   • Efficacy of analgesia by Pain score; will be measured by Numerical Rating Scale (NRS) score (0-10; 0=no pain,1-3=mild,4-6=moderate,7-9=sever,10=most sever) at postoperative12 hours.
2. Secondary outcome measures:

   1. Duration of analgesia, starting from recovery from general anesthesia (GA) to 1st time giving the patient rescue analgesia ( measured by NRS pain score at 0, 6 ,12, 18 and 24 postoperative hours).
   2. Risk of complications from techniques.
   3. Patient satisfaction after surgery
   4. Total intraoperative analgesia dose (fentanyl consumption) and total postoperative analgesia dose (morphine consumption).
   5. Hemodynamics monitoring; measurements of heart rate and mean arterial blood pressure before induction of anesthesia and every 15 minutes during surgery till end of surgery

VII. Statistical analysis:

1. Sample size:

   Sample size calculation was based on pain score after Interscalene block (ISB) in shoulder surgery versus other methods retrieved from previous research (Singelyn et al., 2004) (15). Using G power program version 3.1.9.4 to calculate sample size based on effect size of 0.897 (35 ± 25) versus (13±24), using 2-tailed test, α error =0.05 and power = 80.0%, the total calculated sample size will be 21 in each group at least and by adding 10% to compensate for possible drop out then total sample size per group is 23 cases at least.
2. Statistical analysis:

Data will be analyzed using SPSS (statistical package for social sciences) version 22. Quantitative data will be tested for normality by Kolmogrov-Smironv test then described as mean and standard deviation for normally distributed data, and median and range for non-normally distributed, Qualitative data will be presented as number and percent. The appropriate statistical test will be applied according to data type with the following suggested tests: Student t test and Mann Whitney U test for continuous variables, Chi-Square test for categorical variable.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 to 60,
* ASA classification I or II,
* scheduled for arthroscopic shoulder surgery,
* will be randomized 1:1 into two groups before the induction of general anesthesia (GA)

Exclusion Criteria:

* Patients who refuse participation.
* Have allergies to local anesthetics.
* Phrenic nerve dysfunction.
* Chronic opioid use.
* ASA III or higher classification.
* Coagulopathy.
* Severe chronic obstructive pulmonary disease.
* Local infection at the injection site

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of analgesia | at 12 hours postoperatively
  Will be measured by pain score at 12 hours postoperatively using the Numerical Rating Scale (NRS) (0-10; with 0 means no pain and 10 means most intolerable pain)

SECONDARY OUTCOMES:
Duration of analgesia | Starting from recovery from general anesthesia (GA) to 1st time giving the patient rescue analgesia,
  duration of analgesia measured by Pain score at 0, 6, 12, 18, and 24 hours postoperatively using the Numerical Rating Scale (NRS) 0-10 with 0 means no pain and 10 means most intolerable pain.
Hemodynamics (heart rate) | before induction of anesthesia and every 15 minutes during surgery till end of surgery
  measurements of heart rate (beat per minute)
Total intraoperative analgesic consumption (fentanyl). | During surgery; from induction of anesthesia to end of surgery.
  Need and consumption of fentanyl intraoperatively (ug),
Patient satisfaction | for the first postoperative 24 hours
  very unsatisfied, unsatisfied, neutral, satisfied, very satisfied
Complications of the techniques | From time of injection to the end of first 24 hours postoperative
  Local anesthetics toxicity, pneumothorax, phrenic nerve palsy, hematoma formation
Total postoperative morphine consumption (mg) | From recovery from general anesthesia to end of 24hours postoperatively
  Time to 1st request of rescue analgesia and total dose of postoperative morphine consumption in the studied groups for 24 hours (mg)
Hemodynamics; mean arterial blood pressure (mmHg) | Before induction of anesthesia and every 15 minutes during surgery till end of surgery
  Measurement of mean arterial blood pressure (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Hany Kamal, Prof. of anesthesia and pain, Study Chair — Misr University for Science and Technolog
Locations (1):
- Souad Kafafi University Hospital (SKUH), Faculty of medicine, Misr University for Science and Technology (MUST), Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Demographic Information: Age, sex, race, and other relevant demographic details.
  Baseline Characteristics: Health status, medical history, and any pre-existing conditions prior to the trial.
  Treatment Assignment: Information on the intervention or treatment each participant received.
  Outcome Measures: Data on primary and secondary outcomes as defined in the trial protocol.
  Adverse Events: Reports of any side effects or adverse events experienced by participants during the trial.
  Follow-up Data: Information collected during follow-up periods, including long-term outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 01/06//2025 to 31/5/2026
Access Criteria: Researchers:
  Who: Academic researchers, industry scientists, and regulatory agencies. What: Full IPD, including demographic data, treatment assignments, and outcome measures.
  How: Through data sharing platforms or repositories after submitting a research proposal and obtaining necessary approvals.
  Regulatory Authorities:
  Who: Agencies like the FDA or EMA. What: Full IPD and supporting documentation for oversight and review. How: Direct access during the review process of clinical trial applications.
  Data Sharing Initiatives:
  Who: Collaborating institutions and consortia. What: Aggregated or anonymized IPD for meta-analyses or systematic reviews. How: Via established partnerships and shared databases.
  Public and Patient Advocacy Groups:
  Who: Organizations seeking to promote transparency. What: Summary data and aggregated results, but not individual-level data. How: Through publicly available reports or dashboards.

REFERENCES:
- [Background] Hewson DW, Oldman M, Bedforth NM. Regional anaesthesia for shoulder surgery. BJA Educ. 2019 Apr;19(4):98-104. doi: 10.1016/j.bjae.2018.12.004. Epub 2019 Feb 6. No abstract available. PMID 33456877